CLINICAL TRIAL: NCT05005078
Title: A 16-Week Phase 2a Study of Topical Pirenzepine (WST-057) or Placebo to Treat HIV-Associated Distal Sensory Polyneuropathy (DSP) in Patients With HIV (PWH)
Brief Title: A 16-Week Study of Pirenzepine or Placebo to Treat HIV-Associated Distal Sensory Polyneuropathy in Patients With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WinSanTor, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WST-PZP-004
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: HIV Associated Polyneuropathy
Keywords: Neuropathy; HIV-DSP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: Open label, Part B: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): WST-057 Matching placebo
  Interventions: Drug: Placebo
- WST-057 (Experimental): WST-057 topical solution
  Interventions: Drug: WST-057

INTERVENTIONS:
Drug: WST-057 — WST-057 topical solution
  Arms: WST-057
Drug: Placebo — WST-057 Matching placebo
  Arms: Placebo

SUMMARY:
This is a two-part study of the safety, tolerability, and efficacy of topically administered WST-057 for 16 weeks in subjects with HIV with sensory polyneuropathy.

DETAILED DESCRIPTION:
Phase A: Is an open-labeled feasibility investigation of the safety, tolerability, and limited efficacy in 14 subjects with HIV-associated distal sensory polyneuropathy (HIV-DSP) after topical daily dosing of WST-057 (4% pirenzepine free base monohydrate). Subjects will be stratified based on their baseline scores for pain/discomfort using the Visual Analog Scale (VAS). Subjects will attend visits at screening; Day 0 (baseline); Weeks 4, 8, and 16; and follow-up (Week 18).

Phase B: Is a randomized outpatient, double-blind, placebo-controlled, single-site study of the safety, tolerability, and exploratory efficacy of topically administered WST-057 for 16 weeks in subjects with HIV-associated distal sensory polyneuropathy (HIV-DSP). Stratification of subjects based on baseline pain will be included based on the results of Part A.

Subjects will attend visits at screening; Day 0 (baseline); Weeks 4, 8, and 16; and follow-up (Week 18). Approximately 60 subjects with HIV-DSP will be randomized to 1 of 2 treatment groups in a 3:2 ratio: WST-057 (4 mL) (n = 36 subjects) versus placebo control 4 mL (n = 24 subjects); with the assumption that a total of 50 subjects will complete the study.

This study is designed with 4 periods in both study phases: screening, baseline/day 0, outpatient treatment, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all the following criteria are met:

1. HIV infection documented by serologic testing at screening; virally suppressed on ART.
2. Male and female patients in the age range of 18 to 80 years (inclusive).
3. Diagnosis of HIV-DSP determined by a neurological exam performed by qualified personnel and defined as one or more clinical signs (symmetrical, diminished distal vibration or dull/sharp sensation in feet or reduced ankle reflexes using HNRC CH40);
4. Baseline IENF density <5%ile (ankle) based on age- and sex-adjusted Lauria norms.
5. Provide written informed consent prior to entering the study or undergoing any study procedures.
6. Females should be either not of childbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and must be practicing a highly effective medically acceptable method of contraception, including abstinence; hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device or intrauterine system; or vasectomy (partner), for at least 1 month before the screening visit and for 1 month after the end of the last dose of study drug. If access or use of a highly effective medically acceptable method of contraception is not achievable, then a combination of barrier methods (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge) is acceptable. Eligible female subjects must also have a negative serum beta-human chorionic gonadotropin at the screening visit.
7. Males must use an acceptable form of contraception (e.g., male condom with diaphragm, male condom with cervical cap, or male condom in association with spermicide).
8. If diabetic, glycemic control has been optimized and has been stable for at least three months prior to randomization. Optimal glycemic control (by HgbA1C<7; at discretion of PI) refers to the best possible diabetic control that an individual patient can attain with usual standards of care, which usually takes more than two months to establish.
9. Participating subjects must be reliable, willing, and able to cooperate with all study procedures, including the following:

   * Return for study visits on the required dates
   * Be physically able to inspect calves, tops of ankles, and soles of feet for wounds, infections, or other anomalies, and be able to self-administer the investigational drug to calves and top surface of feet.
   * Be able to accurately and reliably report symptoms (including treatment-emergent signs and symptoms).
   * Take study drug as required by protocol.
10. If diabetic, be on stable antidiabetic treatment (> 2 months prior to screening) (oral or injectable antidiabetic therapy and/or lifestyle) that is not anticipated to change during the course of the study, except if medically required.
11. Be on stable nonpharmacological pain/uncomfortable sensation treatment for at least 4 weeks prior to screening and remain on this stable treatment throughout the study (unless otherwise directed by a physician). Nonpharmacologic pain treatment includes the following: relaxation/hypnosis, physical or occupational therapy, counseling, etc. Episodic or periodic treatments, such as monthly injections for treatment of pain (e.g., local anesthetics) or trans electrical nerve stimulation will not be permitted.
12. Regular and stable use of pharmacological pain/uncomfortable sensation treatment (less than or equal to 30 mg morphine equivalent) for at least 8 weeks prior to screening.
13. General health status must be acceptable for participation in this 16-week clinical study, during screening per judgment of the Investigator. Any question regarding eligibility will be addressed with the medical monitor.
14. Fluency (oral and written) in the language in which the standardized tests will be administered (English or Spanish)

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will be excluded from participating in the study:

1. Current intoxication (BAC > 0.08%) at the screening visit at the discretion of the investigator (breathalyzer analysis).
2. Neuropathy due to exposure to current use/ chemotherapeutic agents or other neurotoxins; at the discretion of the investigator.
3. Individuals with the onset of Type 2 diabetes mellitus before HIV infection.
4. Uncontrolled or Insulin-dependent diabetes mellitus.
5. Proliferative retinopathy or maculopathy requiring acute treatment.
6. Requiring dialysis. Impaired liver function, defined as aspartate aminotransferase or alanineaminotransferase > 3 times the upper limit of normal.
7. Presence of clinically significant peripheral or autonomic neuropathy that is clearly of non HIVN origin.
8. Active and/or systemic infections with hepatitis C (as per investigator judgement following serology results) or syphilis, or a history of severe infection during the 30 days prior to screening.
9. Diagnosis and/or treatment of malignancy (except for basal cell or squamous cell skin cancer, in-situ carcinoma of the cervix, or in-situ prostate cancer) within the past 5 years.
10. Clinically significant diagnosed gastric emptying abnormality (e.g., severe gastroparesis).
11. Clinically significant - urinary retention confirmed by bladder ultrasound regardless of etiology.
12. Uncontrolled glaucoma.
13. Other clinically significant, active (over the past 12 months) disease of the cardiovascular, gastrointestinal, pulmonary, neurological, genitourinary, endocrine, rheumatologic or hematological system that, in the opinion of the Investigator, would compromise the subject's participation in the study, might confound the results of the study, or pose additional risk in administering the study drug.unstable/untreated clinically significant.
14. New treatment with (< 2 months) antioxidant supplements, vitamins, or drugs known to affect oxidative stress and such as Superoxide Dismutase, Alpha Lipoic Acid, Acetyl L-Carnitine and Vitamin B12.
15. Mental incapacity, unwillingness, or language barrier precluding adequate understanding of or cooperation with the study.
16. Women of childbearing potential who are pregnant, breast-feeding, or intend to become pregnant. Women of childbearing potential must have a negative pregnancy test at Screening and must agree to use adequate contraceptive methods during the study and for 1 month after the last dose of study drug (see inclusion criterion 5).
17. History of allergy or sensitivity to M1 antagonists or anticholinergics in general or any of the components of the investigational product formulations.
18. Local (topical) anesthetics or analgesics including lidocaine, capsaicin, cannabinoid (CBD) oil/products or compounded topical pharmaceutical agents.
19. Uncontrolled treated/untreated hypertension (systolic blood pressure [BP] > 180 or diastolic BP > 100 at screening).
20. Amputations of lower extremities or presence of foot ulcers.
21. Clinically significant active macrovascular disease, including myocardial infarction, arrythmias, prolonged QT syndrome, or cerebrovascular event within the past 6 months.
22. A history of severe infection during the 30 days prior to screening.
23. Major surgical procedure during the 90 days prior to screening.
24. History of sensitive skin, as defined by a requirement to use soap and skin products formulated for "sensitive skin," as determined by the Investigator.
25. Currently taking M1 antagonists medicines to treat overactive bladder (anticholinergic agents, such as Gelnique), or antispasmodics.
26. Failure or inability to perform screening or baseline assessments.

    Patients with any condition that could potentially interfere with the conduct of the study or confound efficacy evaluations, including the following as specified in numbers 26 through 32 below:
27. Pain or neuropathy from another cause, as determined by the investigator (including central pain, radiculopathy, painful arthritis, etc.).
28. Active skin or soft-tissue lesions in the dosing area (calves, ankles and tops of feet) affected by neuropathy that are painful or could alter sensation.
29. Exposure to an experimental drug, experimental biologic, or experimental medical device within 3 months before screening.
30. Any open wound(s) and/or sunburn(s) in the dosing area. Subjects who have a wound and/or sunburn at screening that is anticipated to resolve before day -1 can be enrolled.
31. History of a serious skin disease (as determined by the Investigator), such as skin cancer, psoriasis, stasis dermatitis or eczema.
32. Receipt of a tattoo in the dosing area within 12 months of dosing.
33. Known or untreated Lyme disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events as assessed by hematology and clinical pathology blood tests | 16 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by vital signs (blood pressure (diastolic and systolic mmHg), heart rate (beats per minute), respiratory rate (breaths per minute). | 16 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by ECG (measuring p wave, QRS complex, QT interval) | 16 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.
Incidence of Treatment Emergent Adverse Events as assessed by dermal assessment (Draize score 0.0-4.0) score of skin erythema, edema pruritus and dryness score) of the dosing area | 16 weeks
  Safety will be assessed by observing changes in patients' blood tests when compared to normal lab values/ranges after once daily dosing of 1 dose level of WST-057 solution or placebo. The number of participants with treatment-related adverse events as assessed by CTCAEv4.0 will be reported.

SECONDARY OUTCOMES:
IENFD change from baseline for both treated and untreated skin | 16 weeks
  Quantification of IENF density (IENFD) by skin biopsy: This measurement will provide the other co-secondary outcome measures for the study so that effects on both patient function and nerve structure are assessed. IENFD is the gold standard for measuring small fiber neuropathy.
Visual Analogues Score (VAS) for pain assessment | 16 weeks
  Scores are based on self-reported measures of symptoms that are recorded with a single mark placed at one point along a horizontal line 100 mm in length that represents a continuum between the two ends of the scale-"no pain" on the left end of the scale and the "worst imaginable pain" on the right end of the scale.
Neuropathy Total Symptom Score-6 (NTSS-6) | 16 weeks
  The NTSS-6 is a validated tool that assesses intensity and frequency of different pain modalities (aching, burning, prickling & lancinating pain, numbness and allodynia) in patients with neuropathy. Each sensation is reported on a 4-point scale from "Not present" to "Severe." It shows good internal consistency, test-retest reliability, and construct validity.
Medical Outcomes Study HIV Health Survey (MOS-HIV) | 16 weeks
  MOS-HIV is a brief, comprehensive health status measure that has been used extensively in studies of human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS). The 35-item questionnaire includes ten dimensions (health perceptions, pain, physical, role, social and cognitive functioning, mental health, energy, health distress and quality of life (QoL) and takes approximately 5 minutes to complete. Subscales are scored on a 0-100 scale (a higher score indicates better health) and physical and mental health summary scores can be generated.
Patient's Global Impression of Change (PGIC) | 16 weeks
  The PGIC scale will be used to assess patients' perception of changes following treatment (i.e., "feeling better" or "feeling worse"). The PGIC is a 7-point scale from "much improved" to "much worse." The PGIC is commonly used in clinical studies assessing pain relief following treatment, due to its ease of administration and scoring and because it is a generic scale applicable to a wide variety of conditions and treatments including diabetic peripheral neuropathy
Quantitative Sensory Testing (QST) | 16 weeks
  QST for vibration, warm and cold perception thresholds on both great toes will be assessed. A reduction in QST vibration threshold has shown to have high diagnostic value in subjects with HIV-associated neuropathies.
Utah Early Neuropathy Score (UENS) | 16 weeks
  UENS is a simple, rapid, and reproducible test targeted to detect early sensory peripheral neuropathy. It includes motor examination, pin sensation, allodynia, hyperesthesia, large-fiber sensation, and deep tendon reflexes. The sensations are reported on 0-, 1-, or 2-point scoring for normal, reduced or absent vibration or reflexes.
Neuropathic Pain Scale-10 (NPS-10) | 16 weeks
  The NPS-10 will be used to assess the effect of treatments impacting neuropathic pain. It is reported on 0-10 scale with 0 indicating no pain and 10 indicating the most pain imaginable. It is suggested that an NPS-10 score greater than 43 of 100 may indicate the presence of neuropathic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hansen, Study Director — WinSanTor, Inc
Locations (2):
- United States (2):
  - Palmtree Clinical Research, Palm Springs, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No